CLINICAL TRIAL: NCT00951522
Title: A Phase 1 Randomized, Double-Blind, Placebo-Controlled Trial to Assess the Safety, Tolerability, and Pharmacokinetics of GS-9411 in Healthy Male Volunteers
Brief Title: A Trial to Assess the Safety, Tolerability, and Pharmacokinetics of GS-9411 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Thomas O'Riordan, MD, Gilead Sciences, Inc.</
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-221-0102
Record Dates: First submitted 2009-08-03; First posted 2009-08-04 (Estimated); Last update posted 2009-09-25 (Estimated); Status verified 2009-09

CONDITIONS: Cystic Fibrosis; Mucociliary Clearance; Airway Hydration
Keywords: Cystic Fibrosis; CF; Mucociliary Clearance; Epithelial Sodium Channel Inhibitor; ENaC Inhibitor; Airway Hydration; Amiloride
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental): GS-9411 2.4 mg
  Interventions: Drug: GS-9411
- 2 (Experimental): GS-9411 4.8 mg
  Interventions: Drug: GS-9411
- 3 (Experimental): GS-9411 7.2 mg
  Interventions: Drug: GS-9411
- 4 (Experimental): GS-9411 9.6 mg
  Interventions: Drug: GS-9411
- 5 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GS-9411 — Inhaled GS-9411 dissolved in sterile saline
  Arms: 1; 2; 3; 4
Drug: Placebo — Inhaled placebo in sterile saline
  Arms: 5

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of escalating doses of GS-9411 in healthy male volunteers. GS-9411 is a sodium channel inhibitor, that may restore airway hydration and mucociliary clearance in the lung.

DETAILED DESCRIPTION:
GS-9411 is being evaluated as a potential therapy to improve airway hydration and mucociliary clearance in patients with cystic fibrosis. This study is evaluating the safety and tolerability of 4 dose levels of GS-9411 as an inhaled product, compared to a matched placebo.

ELIGIBILITY:
Inclusion Criteria:

* Males 18 to 45 years of age
* No clinically important abnormal physical findings at the screening examination
* No clinically relevant abnormalities in the results of laboratory screening evaluation
* Normal (or abnormal but not clinically significant) ECG
* Normal (or abnormal but not clinically significant) blood pressure (BP) and heart rate(HR).
* Body weight between 70 and 125 kg and body mass index (BMI) between 18 and 28 kg/m2.
* Able to communicate well with the investigator and to comply with the requirements of the entire study.
* Provision of written informed consent to participate as shown by a signature on the volunteer consent form.
* Non-smokers of at least 6 months duration (< 10 pack/year history) prior to study entry.
* Negative for drugs of abuse (including alcohol) at Screening and Day -5.
* Must be willing to abstain from alcohol and strenuous exercise during the 48-hour period prior to admission and during the study.
* Forced expiratory volume in 1 second (FEV1) ≥ 80% of predicted normal for age, gender, and height at Screening and Pre-dose.
* Normal intraocular pressure between 10 and 21 mm Hg.
* Male subjects who are sexually active must be willing to use effective barrier contraception (e.g., condoms) during heterosexual intercourse from Baseline/Day 0 through completion of the study and continuing for at least 90 days from date of last dose of study drug.
* Male subjects must refrain from sperm donation from Day 1 through completion of the study and continuing for at least 90 days from the date of last dose of study drug.

Exclusion Criteria:

* Any prior exposure to GS-9411.
* Administration of any investigational drug in the period 0 to 12 weeks before entry to the study.
* A need for any medication during the period 0 to 5 days before entry to the study, except those deemed by the principal investigator/clinical investigator not to interfere with the outcome of the study.
* Existence of any surgical or medical condition which, in the judgment of the clinical investigator, might interfere with the absorption, distribution, metabolism, or excretion of the drug.
* Presence or history of allergy requiring treatment. Hay fever is allowed unless it is active or has required treatment within the previous 2 months.
* Donation or loss of greater than 400 mL of blood in the period 0 to 12 weeks before entry to the study.
* Serious adverse reaction or hypersensitivity to any drug.
* Presence or history of any pulmonary diseases (e.g., asthma, emphysema, chronic bronchitis, cystic fibrosis, bronchiectasis).
* Consumption of drugs and/or herbal preparations capable of inducing hepatic enzyme metabolism (e.g., barbiturates, rifampicin, carbamazepine, phenytoin, primidone, or St. John's Wort) or enzyme-inhibiting agents (e.g., cimetidine) or similar drugs within 30 days (or 5 half-lives of inducing/inhibiting agent, whichever is longer) of enrollment in this study.
* Major surgery within 6 months of the start of this study.
* Subjects who have experienced a significant upper or lower respiratory tract infection within the 6 weeks prior to admission.
* Subjects with significant history of respiratory, renal, hepatic, cardiovascular (including history of systemic hypertension requiring therapy), metabolic, neurological, hematological, gastrointestinal, cerebrovascular, or other significant medical illness or disorder which, in the judgment of the investigator, may interfere with the study or require treatment which may affect the evaluation of efficacy and safety of the study drug.
* Subjects with elevated liver enzyme concentrations at Screening and at Day -1.
* Hemoglobin level < 130 g/L taken at Screening and at Day -1.
* Serum potassium > 5 mEq/L taken at Screening and at Day -1.
* Poor venous access.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2009-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of 4 escalating doses of GS-9411 in healthy male volunteers | 7 Days

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hodsman, MD, Principal Investigator — Nucleus Network Ltd
Locations (1):
- Nucleus Network, Ltd., Melbourne, Victoria, Australia